CLINICAL TRIAL: NCT01558687
Title: A Multi-center, Open-label, Randomized, Controlled Phase I Trial to Investigate the Effects of Cilengitide (EMD 121974) Using Dynamic MR and FET-PET Imaging as a Pharmacodynamic Measure of Response in Subjects With Newly Diagnosed Glioblastoma
Brief Title: Cilengitide Imaging Trial in Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinuation of development program
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EMR062041-017; 2011-003794-29 (EudraCT Number)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Supratentorial Newly Diagnosed Inoperable Gliobastoma
Keywords: Oncology; newly diagnosed inoperable glioblastoma; temolozomide; radiotherapy; dynamic MRI; Positron emission tomography; [18]FET tracer; cilengitide; World Health Organization [WHO] Grade IV
MeSH Terms: conditions — Neoplasms | interventions — Pharmaceutical Preparations; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A = Cilengitide Group (Experimental): Cilengitide + SoC (Temolozomide + Radiotherapy)
  Interventions: Drug: Drug (including placebo)
- Group B = Control Group (Active Comparator): SoC (Temolozomide + Radiotherapy)
  Interventions: Other: Standard therapy

INTERVENTIONS:
Drug: Drug (including placebo) — Subjects will receive cilengitide monotherapy for 2 weeks (Weeks 1 and 2); thereafter, cilengitide will be given in combination with the standard treatment regimen during Weeks 3 to 36. The standard combination treatment of radiotherapy (RTX) plus Temolozomide (TMZ) will be administered for a maximum of 6 weeks (Weeks 3 to 8), followed by TMZ maintenance treatment starting 4 weeks after RTX (i.e., Week 13) for up to 6 cycles, 4 weeks per cycle.
  Cilengitide monotherapy treatment will be given to subjects in Group A for another 10 months as maintenance treatment (Weeks 37 to 78). Subjects in Group A may continue to receive cilengitide maintenance treatment beyond 10 months (beyond Week 78) until occurrence of progressive disease (PD) or unacceptable toxicity, or withdrawal for any other reason. A 28-day safety follow-up will be performed after the last dose of cilengitide.
  Arms: Group A = Cilengitide Group
Other: Standard therapy — In the first two weeks, treatment of subjects in Group B will be in line with the SoC. Thereafter the standard combination treatment of radiotherapy (RTX) plus Temolozomide (TMZ) will be administered for a maximum of 6 weeks (Weeks 3 to 8), followed by TMZ maintenance treatment starting 4 weeks after RTX (i.e., Week 13) for up to 6 cycles, 4 weeks per cycle.
  Arms: Group B = Control Group

SUMMARY:
The main purpose of this clinical trial is to find out if cilengitide has an effect on brain tumor cells but also particularly on the blood vessels supplying the tumor with nutrient and oxygen in patients newly diagnosed with non-resectable (inoperable) glioblastoma.

In addition, this clinical trial will investigate if the addition of cilengitide in combination with standard treatment prolongs life in patients with non-resectable glioblastoma. Similarly, the duration of response of the cancer to this treatment and the side effects of the therapy will be analyzed. Furthermore, additional data on how the body deals with this substance will be collected (this is called pharmacokinetics or pharmacokinetic (PK) analysis). In this clinical trial the investigators would also like to learn more about the disease and the response to the experimental medication by measuring certain "markers".

This imaging trial will investigate the biological effects of cilengitide monotherapy on the tumor microvascular function and tumor viability in a homogenous non-pretreated subject population with newly diagnosed Gliobastoma (GBM). The purpose of this clinical trial is to study the effect that cilengitide may have on certain markers of cancer in your tumor and/or blood and to learn if there are any disease-related markers that could help in predicting how subjects respond to the administration of cilengitide.

The investigators anticipate that approximately 30 subjects will participate in this clinical trial. The clinical trial will be conducted in approximately 4 medical centers in the following countries: Germany, Poland, and Switzerland. The investigators anticipate the clinical trial will last until the end of 2013. Your participation in the trial may last up to 86 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 to ≤ 70 years at the time of informed consent signature
* Tumor tissue specimens taken from multimodal imaging-guided stereotactic biopsy must be available for histopathological confirmation of GBM and potential subsequent analysis of tissue molecular markers
* Newly diagnosed histologically proven supratentorial GBM (World Health Organization [WHO] Grade IV)
* Subject with non-resectable GBM
* Available dynamic MRI and FET-PET scan prior to randomization
* Available Gd-MRI performed prior randomization
* ECOG Performance status of 0-2
* Stable or decreasing dose of steroids for >= 5 days prior to randomization
* Given written informed consent

Exclusion Criteria:

* Prior chemotherapy within the last 5 years
* Prior RTX of the head (except for low-dose radiotherapy for Tinea capitis)
* Gross total resection/partial resection (GBM surgery), placement of Gliadel® wafer
* Receiving concurrent investigational agents or receipt of an investigational agent within the past 30 days prior to the first day of intensified imaging (W1D1)
* Prior systemic antiangiogenic therapy
* Inability to undergo dynamic MR or FET-PET imaging
* History of allergic reactions attributed to Gadolinium-based contrast agents for MRI, compounds of similar chemical or biological composition
* Planned major surgery for other diseases
* History of recent peptic ulcer disease (endoscopically proven gastric ulcer, duodenal ulcer, or esophageal ulcer) within 6 months prior to enrollment
* History of other malignant disease or acute malignant disease. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for ≥ 5 years are eligible for this study
* Current or history of bleeding disorders and/or history of thromboembolic events
* Clinically manifest myocardial insufficiency (NYHA III, IV) or history of myocardial infarction during the past 6 months prior to enrollment, uncontrolled arterial hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Rate constant for passive contrast agent plasma/interstitium transfer (ktrans) | 2 weeks
  Any change in tumor kinetic model parameter (maximum increase in ktrans) to assess the tumor microvasculature structure and function
Fractional blood plasma volume (vp) | 2 weeks
  Any change in tumor kinetic model parameter (maximum change in vp) to assess the tumor microvasculature structure and function
Maximum tumor to brain ratio (TBRmax) | 2 weeks
  Assessment of tumor amino acid (FET) uptake (tumor viability)

SECONDARY OUTCOMES:
Total tumor volume and enhancing tumor volume | 2 weeks
  Change in total tumor volume and enhancing tumor volume as a measure of the overall level of tumor perfusion during the first 2 weeks of treatment with Cilengitide monotherapy
Interstitial space volume fraction (putative contrast agent distribution volume) (=ve) | 2 weeks
  Change in the tumor extravascular extracellular space volume during the first 2 weeks of treatment with Cilengitide monotherapy
Apparent Diffusion coefficient (ADC) | 2 weeks
  Change in perfusion parameter ADC during the first 2 weeks of treatment with Cilengitide monotherapy
Fractional anisotropy (FA) | 2 weeks
  Change in FA during the first 2 weeks of treatment with Cilengitide monotherapy
Kinetic behavior of [18F]FET uptake | 2 weeks
  Change in tumor amino acid (FET) uptake kinetics during the first 2 weeks of treatment with Cilengitide monotherapy
Mean spin-lattice relaxation time of unbound protons in water | 2 weeks
  Change in Absolute T1(mean spin-lattice relaxation time of unbound protons in water) during the first 2 weeks of treatment with Cilengitide monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ute Klinkhardt, MD, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Merck KGaA Communication Center located in, Darmstadt, Germany